CLINICAL TRIAL: NCT00984308
Title: Diagnosis and Treatment of Sleep Apnea in Cerebrovascular Disease
Acronym: Go To Sleep
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 06-233; NCT00807417 (obsolete NCT alias)
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Results first posted 2015-09-01 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Obstructive Sleep Apnea; Stroke; Transient Ischemic Attack; Hypertension
Keywords: sleep apnea; hypertension; brain ischemia
MeSH Terms: conditions — Sleep Apnea, Obstructive; Stroke; Ischemic Attack, Transient; Hypertension; Sleep Apnea Syndromes; Brain Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group received unattended polysomnography and auto-titrating CPAP if sleep apnea was diagnosed
  Interventions: Procedure: CPAP Therapy for Newly Diagnosed Obstructive Sleep Apnea (OSA)
- Control (Other): The control group received usual clinical care which may include receipt of sleep diagnostic and therapeutic services
  Interventions: Procedure: CPAP Therapy for Newly Diagnosed Obstructive Sleep Apnea (OSA)

INTERVENTIONS:
Procedure: CPAP Therapy for Newly Diagnosed Obstructive Sleep Apnea (OSA) — Continuous Positive Airway Pressure (CPAP) is provided for those patients who are diagnosed with OSA.

SUMMARY:
Sleep apnea is common among Veterans with cerebrovascular disease (stroke or transient ischemic attack [TIA]), leads to hypertension, and is associated with recurrent stroke and death. Although continuous positive airway pressure (CPAP) safely treats sleep apnea, few Veterans with cerebrovascular disease are diagnosed with sleep apnea or offered treatment.

DETAILED DESCRIPTION:
The project sought to evaluate whether a diagnostic and therapeutic intervention strategy among Veterans with cerebrovascular disease and hypertension using unattended polysomnography and auto-titrating CPAP with a targeted adherence evaluation and educational protocol resulted in: an improved rate of diagnosed sleep apnea, an improved rate of treated sleep apnea, and improved blood pressure control.

ELIGIBILITY:
Inclusion Criteria:

Stroke or Transient Ischemic Attack Hypertension

Exclusion Criteria:

* Prior diagnosis of sleep apnea or other sleep disorder
* Life expectancy < 6 months or Hospice
* Non-English speaker
* Unable/unwilling to use mask
* Inability to give informed consent
* Oxygen dependent COPD
* Chronic renal failure with dialysis
* Active Suicidal Ideation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2008-12-23 (Actual); Primary Completion 2011-09-30 (Actual); Study Completion 2011-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn M. Bravata, MD, Principal Investigator — Richard L. Roudebush VA Medical Center, Indianapolis, IN
Locations (2):
- United States (2):
  - VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut
  - Richard L. Roudebush VA Medical Center, Indianapolis, IN, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Roger VL, Go AS, Lloyd-Jones DM, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Soliman EZ, Sorlie PD, Sotoodehnia N, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2012 update: a report from the American Heart Association. Circulation. 2012 Jan 3;125(1):e2-e220. doi: 10.1161/CIR.0b013e31823ac046. Epub 2011 Dec 15. No abstract available. PMID 22179539
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Executive summary: heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):143-52. doi: 10.1161/CIR.0b013e318282ab8f. No abstract available. PMID 23283859
- [Background] Go AS, Mozaffarian D, Roger VL, Benjamin EJ, Berry JD, Borden WB, Bravata DM, Dai S, Ford ES, Fox CS, Franco S, Fullerton HJ, Gillespie C, Hailpern SM, Heit JA, Howard VJ, Huffman MD, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Magid D, Marcus GM, Marelli A, Matchar DB, McGuire DK, Mohler ER, Moy CS, Mussolino ME, Nichol G, Paynter NP, Schreiner PJ, Sorlie PD, Stein J, Turan TN, Virani SS, Wong ND, Woo D, Turner MB; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2013 update: a report from the American Heart Association. Circulation. 2013 Jan 1;127(1):e6-e245. doi: 10.1161/CIR.0b013e31828124ad. Epub 2012 Dec 12. No abstract available. PMID 23239837
- [Result] Sico JJ, Phipps MS, Yaggi HK, Burrus N, Ferguson J, McClain V, Austin C, Li X, Bravata DM. Ambulatory blood pressure monitoring among patients with cerebrovascular disease. Blood Press Monit. 2011 Oct;16(5):211-7. doi: 10.1097/MBP.0b013e32834b4d6c. PMID 21885958
- [Result] Bravata DM, Ferguson J, Miech EJ, Agarwal R, McClain V, Austin C, Struve F, Foresman B, Li X, Wang Z, Williams LS, Dallas MI, Couch CD, Sico J, Fragoso C, Matthias MS, Chumbler N, Myers J, Burrus N, Dube A, French DD, Schmid AA, Concato J, Yaggi HK. Diagnosis and Treatment of Sleep Apnea in patients' homes: the rationale and methods of the "GoToSleep" randomized-controlled trial. J Clin Sleep Med. 2012 Feb 15;8(1):27-35. doi: 10.5664/jcsm.1654. PMID 22334806
- [Result] Schmid AA, Yaggi HK, Burrus N, McClain V, Austin C, Ferguson J, Fragoso C, Sico JJ, Miech EJ, Matthias MS, Williams LS, Bravata DM. Circumstances and consequences of falls among people with chronic stroke. J Rehabil Res Dev. 2013;50(9):1277-86. doi: 10.1682/JRRD.2012.11.0215. PMID 24458967
- [Result] Zis P, Spengos K, Manios E, Vemmos K, Zis V, Dimopoulos MA, Zakopoulos N. Ambulatory blood pressure monitoring in acute stroke: the importance of time rate of blood pressure variation. Blood Press Monit. 2012 Oct;17(5):220-1; author reply 221-2. doi: 10.1097/MBP.0b013e3283588e8a. No abstract available. PMID 22968110

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Control
Started | 110 | 115
Completed | 92 | 109
Not Completed | 18 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 110 | 115 | 225
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.4) | 70.2 (10.1) | 70 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 6
  Male | 109 | 110 | 219

OUTCOME MEASURES:

1. Primary Outcome: Sleep Apnea Diagnosis Rate
Description: The number of patients with a diagnosis of sleep apnea
Time Frame: The entire study period (baseline and up to one-year)
Population: The intervention patients had polysomnography at baseline (n=102) whereas control patients either had polysomnography as part of usual care (n=7) or at the end of the study as part of the study protocol (n=85). The n=7 patients who had polysomnography as part of usual care were included in the analysis for this outcome.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 102 | 7
participants | 58 | 5

2. Primary Outcome: Hypertension Control
Description: Medication-Adjusted Systolic Blood Pressure
Time Frame: One year
Population: ITT
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 110 | 115
mm Hg | 157.4 (25) | 161.6 (24.3)

3. Secondary Outcome: Sleep Apnea Treatment Rate
Time Frame: One year
Population: Among the 58 intervention patients with a diagnosis of sleep apnea, CPAP data were available for 57. Among the 7 control patients who received polysomnography as part of usual care, 5 had sleep apnea: CPAP data were available for 4 patients (2 did not receive any CPAP and 2 had CPAP therapy), the data card was unavailable for 1 patient.
Measure: Number; unit: participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 57 | 2
participants | 22 | 0

ADVERSE EVENTS:
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 5/110 | 2/115
Other Adverse Events (participants affected / at risk) | 22/110 | 30/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=110) | Control (N=115)
stroke (Nervous system disorders) | 0 (0) | 1 (1) — new stroke event in patient with history of cerebrovascular disease
Transient ischemic attack (TIA) (Nervous system disorders) | 1 (1) | 1 (1)
Congestive heart failure (CHF) (Cardiac disorders) | 3 (3) | 0 (0)
Acute myocardial infarction (AMI) (Cardiac disorders) | 0 (0) | 0 (0)
DEATH (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=110) | Control (N=115)
Falls (General disorders) | 22 (22) | 30 (30)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes